CLINICAL TRIAL: NCT01170247
Title: Intranasal Ketamine Versus Intramuscular Ketamine for Procedural Sedation: A Prospective Randomized, Double-blinded, Placebo Controlled Study
Brief Title: Intranasal Ketamine Versus Intramuscular Ketamine for Procedural Sedation in Pediatric Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: lack of enrollment
Sponsor: University of Iowa (Other)
Responsible Party: Principal Investigator, Brett A Faine, Clinical Pharmacy Specialist, University of Iowa
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201006786; University of Iowa
Record Dates: First submitted 2010-07-21; First posted 2010-07-27 (Estimated); Results first posted 2017-07-02 (Actual); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Sedation
Keywords: Procedural Sedation
MeSH Terms: interventions — Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intranasal Ketamine (Experimental)
  Interventions: Drug: Ketamine
- Intramuscular Ketamine (Active Comparator)
  Interventions: Drug: Ketamine

INTERVENTIONS:
Drug: Ketamine — Intranasal Ketamine (100 mg/mL)
  Arms: Intranasal Ketamine
Drug: Ketamine — Intramuscular Ketamine
  Arms: Intramuscular Ketamine

SUMMARY:
The purpose of this study is to determine if intranasal ketamine is equally as effective and safe as intramuscular ketamine for procedural sedation in pediatric patients.

ELIGIBILITY:
Inclusion Criteria:

* pediatric patients age 2 to 17 years old
* have a laceration of 4 cm on the face or 7 cm on the remainder of the body
* Require procedural sedation to repair the laceration

Exclusion Criteria:

* Patients with abnormal nasal physiology which would not allow for adequate medication delivery
* Unable to have a guardian present to consent on their behalf
* Allergy to ketamine
* Significant cardiac history (myocardial ischemia, heart failure, arrhythmias)
* Presenting with a head injury associated with possible intracranial hypertension
* Pregnancy
* Lacerations that require repair from a consult service

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2011-01; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hogrefe, MD, Principal Investigator — University of Iowa; Brett Faine, Pharm.D., Principal Investigator — University of Iowa; Andrew Nugent, MD, Principal Investigator — University of Iowa
Locations (1):
- University of Iowa Hospitals and Clinics, Iowa City, Iowa, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 6 months
Groups:
- Intranasal Ketamine: Enrolled 2 patients over 6 month period
Period: Overall Study
Arm/Group | Intranasal Ketamine | Intramuscular Ketamine
Started | 2 | 1
Completed | 2 | 1
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intranasal Ketamine | Intramuscular Ketamine | Total
Number analyzed (Participants) | 2 | 1 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 3 (1) | 3 (NA) — Standard deviation not calculated for one patient | 3 (0)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 2 | 0 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 1 | 3
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 2 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Onset of Sedation
Description: Minutes it takes until the patient is cooperative enough for the procedure
Time Frame: Every 60 seconds through study completion
Measure: Count of Participants; unit: Participants
Arm/Group | Intranasal Ketamine | Intramuscular Ketamine
Number analyzed (Participants) | 2 | 1
Participants | NA — Data not collected | NA — Data not collected

ADVERSE EVENTS:
Groups:
- Intranasal Ketamine: None Reported
- Intramuscular Ketamine: None report
Arm/Group | Intranasal Ketamine | Intramuscular Ketamine
Serious Adverse Events (participants affected / at risk) | 0/2 | 0/1
Other Adverse Events (participants affected / at risk) | 0/2 | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No